CLINICAL TRIAL: NCT04682106
Title: A Multiple-Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of an LY3493269 Formulation in Healthy Participants
Brief Title: A Study of LY3493269 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17552; J1X-MC-GZHF (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-12-22; First posted 2020-12-23 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Healthy
MeSH Terms: interventions — N-(8-(2-hydroxybenzoyl)amino)caprylate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Placebo (Placebo Comparator): Participants received placebo orally once daily (QD) for three consecutive days.
  Interventions: Drug: Placebo
- 8 Milligrams (mg) LY3493269 + 600 mg Salcaprozate Sodium (SNAC) (Experimental): Participants received 8 mg LY3493269 and 600 mg SNAC QD administered orally for three consecutive days.
  Interventions: Drug: LY3493269; Drug: Salcaprozate Sodium
- 24 mg LY3493269 + 600 mg SNAC (Experimental): Participants received 24 mg LY3493269 and 600 mg SNAC QD administered orally for three consecutive days.
  Interventions: Drug: LY3493269; Drug: Salcaprozate Sodium
- 12 mg LY3493269 + 300 mg SNAC (Experimental): Participants received 12 mg LY3493269 and 300 mg SNAC QD administered orally for three consecutive days.
  Interventions: Drug: LY3493269; Drug: Salcaprozate Sodium
- 4 mg LY3493269 + 300 mg SNAC (Experimental): Participants received 4 mg LY3493269 and 300 mg SNAC QD administered orally for three consecutive days.
  Interventions: Drug: LY3493269; Drug: Salcaprozate Sodium

INTERVENTIONS:
Drug: LY3493269 — Administered orally.
  Arms: 12 mg LY3493269 + 300 mg SNAC; 24 mg LY3493269 + 600 mg SNAC; 4 mg LY3493269 + 300 mg SNAC; 8 Milligrams (mg) LY3493269 + 600 mg Salcaprozate Sodium (SNAC)
Drug: Placebo — Administered orally.
  Arms: Placebo
Drug: Salcaprozate Sodium — Administered orally.
  Arms: 12 mg LY3493269 + 300 mg SNAC; 24 mg LY3493269 + 600 mg SNAC; 4 mg LY3493269 + 300 mg SNAC; 8 Milligrams (mg) LY3493269 + 600 mg Salcaprozate Sodium (SNAC)

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of LY3493269 in healthy participants. The blood tests will be performed to check how much LY3493269 gets into the bloodstream, how long the body takes to eliminate it and how body handles LY3493269. The study will last up to approximately 71 days for each participant, including screening

ELIGIBILITY:
Inclusion Criteria:

1. Are male or female not of childbearing potential
2. Body mass index within the range of 19.0 to 40.0 kilograms per square meter (kg/m²) (inclusive)
3. Participants who are healthy as determined through medical evaluation including screening medical history, physical examination, vital signs, clinical laboratory tests, and electrocardiogram (ECG)
4. Have clinical laboratory test results within normal reference range for the population or clinical research unit (CRU), or results with acceptable deviations that are judged to be not clinically significant by the investigator
5. Have venous access sufficient to allow blood sampling as per the protocol.

Exclusion Criteria:

1. Have a significant history of or current CV (for example, myocardial infarction, congestive heart failure, cerebrovascular accident, venous thromboembolism, etc.), respiratory, renal, GI, endocrine, hematological (including history of thrombocytopenia), or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk while taking the IP; or of interfering with the interpretation of data
2. Have undergone any form of bariatric surgery
3. Have a history of gastrointestinal (GI) bleeding or duodenal ulcers
4. Have a personal or family history of medullary thyroid carcinoma or have multiple endocrine neoplasia syndrome type 2
5. Have a history of acute or chronic pancreatitis, or elevation in serum lipase and/or amylase levels greater than 1.5 times the upper limit of normal (ULN)
6. Have clinical signs or symptoms of liver disease, acute or chronic hepatitis
7. Have evidence of significant active neuropsychiatric disease as determined by the investigator
8. Have been treated with prescription drugs that promote weight loss within 3 months prior to screening
9. Are currently enrolled in a clinical study involving an IP or any other type of medical research judged not to be scientifically or medically compatible with this study
10. Have participated within the past 30 days of screening in a clinical study involving an investigational product (IP); at least 5 half-lives or 30 days, whichever is longer, should have passed
11. Have an abnormality in the 12-lead ECG at screening that, in the opinion of the investigator, increases the risks associated with participating in the study or may confound ECG (QT) data analysis, such as a QTcF greater than (>) 450 milliseconds (msec) for males and > 470 msec for females, short PR interval (< 120 msec), or PR interval > 220 msec, second and third atrioventricular block, intraventricular conduction delay with QRS >120 msec, right bundle branch block, left bundle branch block or Wolff-Parkinson-White syndrome
12. Have serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 times (X) ULN or total bilirubin level (TBL) >1.5X ULN
13. Show evidence of HIV infection and/or positive human HIV antibodies
14. Show evidence of hepatitis C and/or positive hepatitis C antibody
15. Show evidence of hepatitis B, positive hepatitis B core antibody, and/or positive hepatitis B surface antigen
16. Have donated blood of more than 450 mL, or have participated in a clinical study that required similar blood volume drawn within the past 3 calendar months
17. Have known allergies to LY3493269, related compounds, or any components of the formulation (including SNAC), or a history of significant atopy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | 8 Milligrams (mg) LY3493269 + 600 mg Salcaprozate Sodium (SNAC) | 24 mg LY3493269 + 600 mg SNAC | 12 mg LY3493269 + 300 mg SNAC | 4 mg LY3493269 + 300 mg SNAC
Started | 8 | 8 | 8 | 8 | 8
Received at Least One Dose of Study Drug | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug.
Groups:
- Placebo: Participants received placebo orally QD for three consecutive days.
- 8 mg LY3493269 + 600 mg SNAC: Participants received 8 mg LY3493269 and 600 mg SNAC QD administered orally for three consecutive days.
- Total: Total of all reporting groups
Arm/Group | Placebo | 8 mg LY3493269 + 600 mg SNAC | 24 mg LY3493269 + 600 mg SNAC | 12 mg LY3493269 + 300 mg SNAC | 4 mg LY3493269 + 300 mg SNAC | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.9 (8.7) | 39.1 (9.9) | 45.5 (10.3) | 44.4 (6.7) | 45.9 (7.0) | 44.0 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 0 | 1
  Male | 8 | 8 | 8 | 7 | 8 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 8 | 8 | 8 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 8 | 8 | 8 | 8 | 8 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 8 | 8 | 8 | 8 | 8 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Treatment-Emergent Adverse Event(s) (TEAEs)
Description: TEAE is an untoward medical occurrence that emerges during a defined treatment period, having been absent pretreatment, or worsens relative to the pretreatment state, and does not necessarily have to have a causal relationship with this treatment.
  A summary of serious adverse events (SAEs), TEAEs and other non-serious adverse events (AEs), regardless of causality, were reported in the Adverse Events section of this record.
Time Frame: Baseline through Day 44
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | 8 mg LY3493269 + 600 mg SNAC | 24 mg LY3493269 + 600 mg SNAC | 12 mg LY3493269 + 300 mg SNAC | 4 mg LY3493269 + 300 mg SNAC
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
Participants | 4 | 8 | 8 | 7 | 6

2. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to 24 Hours (AUC [0-24]) of LY3493269
Description: PK: AUC (0-24) of LY3493269
Time Frame: Day 3: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, & 24 hours post dose
Population: All enrolled participants who received at least one dose of LY3493269 and had at least one evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Groups:
- 8 mg LY3493269 + 600 mg SNAC: Participants received consecutive once-daily oral doses of 8 mg LY3493269 and 600 mg SNAC QD administered orally for three consecutive days.
- 24 mg LY3493269 + 600 mg SNAC: Participants received consecutive once-daily oral doses of 24 mg LY3493269 and 600 mg SNAC QD administered orally for three consecutive days.
- 12 mg LY3493269 + 300 mg SNAC: Participants received consecutive once-daily oral doses of 12 mg LY3493269 and 300 mg SNAC QD administered orally for three consecutive days.
- 4 mg LY3493269 + 300 mg SNAC: Participants received consecutive once-daily oral doses of 4 mg LY3493269 and 300 mg SNAC QD administered orally for three consecutive days.
Arm/Group | 8 mg LY3493269 + 600 mg SNAC | 24 mg LY3493269 + 600 mg SNAC | 12 mg LY3493269 + 300 mg SNAC | 4 mg LY3493269 + 300 mg SNAC
Number analyzed (Participants) | 8 | 7 | 7 | 8
nanograms*hours per milliliter (ng*h/mL) | 2960 (137) | 9680 (46) | 4850 (146) | 1150 (77)

3. Secondary Outcome: PK: Maximum Concentration (Cmax) of LY3493269
Description: PK: Cmax of LY3493269
Time Frame: Day 3: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, & 24 hours post dose
Population: All enrolled participants who received at least one dose of LY3493269 and had at least one evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 8 mg LY3493269 + 600 mg SNAC | 24 mg LY3493269 + 600 mg SNAC | 12 mg LY3493269 + 300 mg SNAC | 4 mg LY3493269 + 300 mg SNAC
Number analyzed (Participants) | 8 | 7 | 7 | 8
nanogram per milliliter (ng/mL) | 166 (137) | 527 (44) | 270 (122) | 62.6 (84)

ADVERSE EVENTS:
Time Frame: Baseline to 44 Days
Description: All enrolled participants who received at least one dose of study drug. Participants were analyzed based on the actual treatment they received.
Arm/Group | Placebo | 8 mg LY3493269 + 600 mg SNAC | 24 mg LY3493269 + 600 mg SNAC | 12 mg LY3493269 + 300 mg SNAC | 4 mg LY3493269 + 300 mg SNAC
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/8 | 8/8 | 8/8 | 7/8 | 6/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | 8 mg LY3493269 + 600 mg SNAC (N=8) | 24 mg LY3493269 + 600 mg SNAC (N=8) | 12 mg LY3493269 + 300 mg SNAC (N=8) | 4 mg LY3493269 + 300 mg SNAC (N=8)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 5 (5) | 1 (1) | 4 (4) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (6) | 3 (5) | 4 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (11) | 5 (7) | 3 (39) | 0 (0)
Catheter site bruise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Catheter site erythema (General disorders) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 2 (2)
Catheter site pain (General disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Medical device site erythema (General disorders) | 2 (3) | 6 (8) | 2 (2) | 2 (3) | 0 (0)
Medical device site laceration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Medical device site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ulcer (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (6) | 7 (8) | 6 (6) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (5) | 2 (2) | 3 (4) | 1 (3)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-03-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT04682106/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/06/NCT04682106/SAP_001.pdf